CLINICAL TRIAL: NCT05703906
Title: Teleneurorehabilitation for the Continuity of Care Post-stroke: a Multicentric Pilot Study
Acronym: TELEICTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: IRCCS Centro Neurolesi Bonino Pulejo (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Fondazione Mondino (Other); IRCCS San Raffaele Roma (Other); Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017.16
Record Dates: First submitted 2022-12-12; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2022-12

CONDITIONS: Stroke
Keywords: Stroke; Telerehabilitation; Feasibility; Virtual reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (Experimental): All patients will receive a kit home-based consisting of a tablet home, an exercise equipment and access to a daily individualized training program based on their needs (i.e., motor, language and/or cognitive training programs).
  The exercise program and patients' sessions will be remotely supervised by therapists.
  Interventions: Behavioral: Telerehabilitation - VRRS Khymeia

INTERVENTIONS:
Behavioral: Telerehabilitation - VRRS Khymeia — Participants will receive an individualized, multidomain exercise program set up by the therapist, based on their needs. The intervention applied will consist of 20 sessions of motor, language and/or cognitive training distributed in five sessions for week, each lasting 1 hour. Remotely, the therapist will supervise the participant's exercise program.

SUMMARY:
The main aim of this longitudinal, pilot study is to evaluate the feasibility of a multi-domain (i.e., motor, language and cognitive domains) telerehabilitation system using the Virtual Reality Rehabilitation System (VRRS, Khymeia) in patients with stroke. Furthermore, data on patients' needs and clinical data will be collected before and after treatment and then analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Single ischemic stroke documented by CT/ MRI;
* 2 to 18 months after the event.

Exclusion Criteria:

* medical history or presence of cognitive decline (MoCA<17.54)
* recent fractures
* History of mental disorders (major depression, psychosis)
* History/presence of other neurological disorders that may interfere with outcome
* Presence of other internal pathologies that may interfere with outcome or treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of telerehabilitation system | 6 weeks
  Feasibility will be measured by calculating the adherence to treatment (i.e. percentage of training sessions completed).
Feasibility of telerehabilitation system | 6 weeks
  Feasibility will be measured with the Technology Acceptance Model (TAM), a specific questionnaire used to quantify the likelihood of technology acceptance, consisting of 12 items, six assessing perceived usefulness and six assessing perceived ease of use.
Feasibility of telerehabilitation system | 6 weeks
  Feasibility will be measured with the System Usability Questionnaire (SUS), a 10 item questionnaire with five response options: from Strongly agree to Strongly disagree.

SECONDARY OUTCOMES:
Change in measure of quality of life | Baseline up to 6 weeks
  Quality of life will be measured by the Short-Form-36 Health Survey (SF-36), a questionnaire comprising 36 questions that cover 8 domains of health. Each of the 8 summed scores is linearly transformed onto a scale from 0 (negative health) to 100 (positive health) to provide a score for each domain. Each domain can be used independently.
Change in measure of quality of life | Baseline up to 6 weeks
  Quality of life will be measured by the EuroQol-5 dimensions (EQ-5D), a questionnaire measuring 5 dimensions described by 3 possible levels of problems (i.e., none, mild-to-moderate, severe). Respondent's answers are translated into a preference-based score, yielding an index score based on a scale from 0.000 (death) to 1.000 (perfect health). The 5 dimensions can be converted to a single utility value (EQ-Index score).
Change in motor functions | Baseline up to 6 weeks
  Change in motor functions will be assessed with the Fugl-Meyer Assessment (FMA), a stroke-specific scale which assesses the motor functioning in patients with post-stroke. There are 3 values for each of the 5 domain: 0 (severe impairment), 1 (moderate impairment), 2 (preserved function). The 5 domains assessed include: motor function (upper limb maximum score = 66; lower limb maximum score = 34), sensory function (maximum score = 24), balance (maximum score = 14), joint range of motion (maximum score = 44), joint pain (maximum score = 44), for an overall maximum score of 226 points.
Change in motor functions | Baseline up to 6 weeks
  Assessed with the Nine hole pegboard test (NHPT), to measure finger dexterity. It is administered by asking the participant to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. Scores are based on the time taken to complete the activity, recorded in seconds.
Change in motor functions | Baseline up to 6 weeks
  Assessed with the Box and block test (BBT). The patient has to carry as much cubes as possible, one by one, from a container to another one in one minute. The test is performed with both hands.
Change in motor functions | Baseline up to 6 weeks
  Assessed with the Ashworth Spasticity Scale. The therapist evaluates the spasticity of the muscles. There are 5 values: 0 (no increase in muscle tone), 1 (slight increase in muscle tone), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone), 4 (affected part rigid in flexion or extension).
Change in linguistic functions | Baseline up to 6 weeks
  Aachen Aphasie Test (AAT)
Change in cognitive functions | Baseline up to 6 weeks
  Assessed with the Montreal Cognitive Assessment (MoCA), a cognitive screening tool comprising 16 items and 11 categories to assess multiple cognitive domains. The total possible score is 30, corresponding to a good performance.
Change in cognitive functions | Baseline up to 6 weeks
  Assessed with the Bells test, a cancellation test that allows for a quantitative and qualitative assessment of visual neglect in the near extra personal space. The total number of cancelled bells is recorded as well as the time taken to complete. The maximum score is 35.
Change in cognitive functions | Baseline up to 6 weeks
  Assessed with the verbal fluency test. Participants have to produce as many words as possible from a semantic and a phonemic category in 1 minute.
Change in Independence (Activities of Daily Living) | Baseline up to 6 weeks
  Assessed with the Barthel Index (BI). It comprises 10 ADL/mobility activities, items are rated based on the amount of assistance required to complete each activity. Each item score ranges from 0 (dependent) to 10 (independent).
Change in behavior (depression) | Baseline up to 6 weeks
  Assessed with the Beck Depression Inventory (BDI). Items are on a four-point scale that ranges from 0 to 3. Ratings are summed to provide a total score ranging from 0-63. Scores >10 generally meet the threshold for a diagnosis of depression.
Change in caregiver burden | Baseline up to 6 weeks
  Assessed with the Zarit Burden Interview (ZBI). It comprises 22 items with a score ranging from 0 ("never" to 4 ("nearly always"). Total scores are obrained by summing all items endorsed.
Satisfaction of the treatment | 6 weeks
  Client Satisfaction Questionnaire, it consists of a 6 item questionnaire with five response options: from 0 to 4, where 0 reflects a negative response and 4 reflects a positive response.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Cacciante, MSc, Principal Investigator — IRCCS San Camillo Hospital
Locations (1):
- IRCCS San Camillo Hospital, Venice, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cacciante L, Kiper P, Garzon M, Baldan F, Federico S, Turolla A, Agostini M. Telerehabilitation for people with aphasia: A systematic review and meta-analysis. J Commun Disord. 2021 Jul-Aug;92:106111. doi: 10.1016/j.jcomdis.2021.106111. Epub 2021 May 13. PMID 34052617
- [Background] Cacciante L, Pieta CD, Rutkowski S, Cieslik B, Szczepanska-Gieracha J, Agostini M, Kiper P. Cognitive telerehabilitation in neurological patients: systematic review and meta-analysis. Neurol Sci. 2022 Feb;43(2):847-862. doi: 10.1007/s10072-021-05770-6. Epub 2021 Nov 25. PMID 34822030